CLINICAL TRIAL: NCT00748111
Title: Thrombus and Inflammation in Sudden Cardiac DEath
Brief Title: Thrombus and Inflammation Study in Sudden Cardiac DEath
Acronym: TIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P080201
Record Dates: First submitted 2008-07-31; First posted 2008-09-08 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Sudden Cardiac Death; Acute Myocardial Infarction
Keywords: Sudden death; Out of hospital cardiac arrest; Acute myocardial infarction; Acute coronary syndrome
MeSH Terms: conditions — Death, Sudden, Cardiac; Death, Sudden; Out-of-Hospital Cardiac Arrest; Acute Coronary Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Sudden cardiac death hospitalized
  Interventions: Other: Blood sample
- 2 (Experimental): Acute myocardial infarction
  Interventions: Other: Blood sample
- 3 (Experimental): Angioplasty procedures programmed
  Interventions: Other: Blood sample
- 4 (Experimental): Sudden cardiac death hospitalized without coronary syndrome
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Blood sample and thrombus sample

SUMMARY:
Sudden death is a natural death occurring within one hour after the onset of symptoms. It remains a major public health problem and accounts for 5 to 10 % of the annual total mortality ie about 300.000 in the United States. Despite community-based interventions, overall survival remains below 5%. Better understanding of the mechanisms causing sudden death could allow early identification of high risk subjects and implementation of specific prevention strategies. The cause of more than 90% of sudden deaths is cardiac with ventricular fibrillation or fast ventricular tachycardia complicating an underlying heart disease. Coronary heart disease and its consequences account for at least 80% of sudden cardiac deaths. Several risk factors associated with sudden death and not with myocardial infarction have been identified in population-based studies. However, the relationship between the occurrence of a coronary artery occlusion and the onset of arrhythmia is unclear. In particular, coronary artery occlusion can be rapidly followed by chest pain, which acts as a signal and allows identification of patients for emergency reperfusion. However, in some cases, the coronary artery occlusion is followed by a sudden onset of arrhythmia and sudden death. Recent data suggest that acute coronary occlusion is caused by plaque erosion or rupture and is followed by an intense local inflammation and rapid thrombus formation. Our hypothesis is that the speed of thrombus formation and coronary occlusion determines the clinical symptoms. Slow and progressive thrombus formation is likely to induce myocardial pre-conditioning thereby reducing the occurrence of ventricular arrhythmia. In contrast, rapid thrombus formation followed by acute coronary artery occlusion and ischemia is more likely to trigger fatal ventricular arrhythmia. During angioplasty procedures, coronary artery thrombus are aspirated, providing the opportunity for pathological studies. The aim of the TIDE study (Thrombus and Inflammation in Sudden Death) is therefore to compare the composition and age of thrombus collected at the site of coronary occlusion in patients with sudden death due to acute coronary artery occlusion and patients with an acute myocardial infarction without ventricular arrhythmia. The following hypothesis will be tested : fresh thrombus is more frequent in patients with sudden cardiac death versus patients with acute myocardial infarction without ventricular arrhythmia.

DETAILED DESCRIPTION:
Sudden death is a natural death occurring within one hour after the onset of symptoms. It remains a major public health problem and accounts for 5 to 10 % of the annual total mortality ie about 40 000 deaths in France and 300.000 in the United States.(1) Despite community-based interventions, overall survival remains below 5%. (2) Better understanding of the mechanisms causing sudden death could allow early identification of high risk subjects and implementation of specific prevention strategies. (3)The cause of more than 90% of sudden deaths is cardiac with ventricular fibrillation or fast ventricular tachycardia complicating an underlying heart disease. (4) Coronary heart disease and its consequences account for at least 80% of sudden cardiac deaths and hypertrophic and dilated cardiomyopathies account for another 10 to 15% of cardiac causes.(4,5) Several risk factors associated with sudden death and not with myocardial infarction have been identified in population-based studies.(6-10) However, the relationship between the occurrence of a coronary artery occlusion and the onset of arrhythmia is unclear.The Framingham study reported that sudden death occurred without prior manifestations of coronary heart disease in more than 50% of men and 65% of women. (11) Data from 10 countries from WHO MONICA PROJECT show that sudden deaths are more frequent than non sudden coronary deaths until age 60. (figure). In a study on the value of immediate coronary angiography and angioplasty in survivors of SCD, a recent coronary artery occlusion was found in over 50% of patients and unstable coronary artery lesions in 20% (12). In two series based on autopsies, the rate of coronary artery lesions in non-survivors of SCD was over 80% (13-15). In a study based on autopsies of non-survivors of SCD, fresh thrombus was found in a majority of cases. (2)Furthermore, noninflammatory plaque erosion was found as an underlying cause to thrombus formation in 40% of cases (14). In this case, thrombus is formed on a denuded endothelial plaque surface and is in direct contact with activated smooth muscle cells. In 211 patients with non-complicated acute myocardial infarction caused by acute coronary occlusion, SASKIA et al studied the age of intracoronary thrombi, aspirated during angioplasty (16). In at least 50% of patients, thrombi were days or weeks old, thereby suggesting ischemic pre-conditioning in this sub-group of acute myocardial infarction patients with no ventricular arrhythmia. Maier et al studied intra-coronary concentrations of selected inflammatory biomarkers in 42 patients with acute myocardial infarction (17). High levels of interleukin 6 and serum amyloid A were found at the occlusion site; and these levels were even higher in patients with no previous clinical symptoms before the acute myocardial infarction. These data suggest that plaque erosion or rupture is followed by an intense local inflammation and rapid thrombus formation. Our hypothesis is that the speed of thrombus formation and coronary occlusion determines the clinical symptoms. Slow and progressive thrombus formation is likely to induce myocardial pre-conditioning thereby reducing the occurrence of ventricular arrhythmia. In contrast, rapid thrombus formation followed by acute coronary artery occlusion and ischemia is more likely to trigger fatal ventricular arrhythmia. We also believe that a precise determination of endothelial cell apoptosis, plaque erosion, and systemic and local inflammation could shed light on the pathogenic mechanisms prevailing in SCD due to acute coronary artery occlusion. Protection and thrombectomy devices were recently developed to avoid distal embolisation during angioplasty procedures in saphenous vein graphs or during angioplasty for acute myocardial infarction. These devices provide the unique opportunity to harvest blood and thrombi from the site of coronary occlusion. The aspirate can be used to study the speed and the intensity of local thrombus formation. The use of such techniques could be extended to patients with a SCD due to an acute coronary artery occlusion and the data compared to that of patients with an acute myocardial infarction without ventricular arrhythmia. Furthermore, markers of endothelial cell apoptosis, local and systemic inflammatory biomarkers in the culprit coronary artery and in the systemic blood could be studied in such patients and also during angioplasty procedures performed in patients with stable coronary lesions.(18-23) The aim of the TIDE study (Thrombus and Inflammation in Sudden Death) is therefore to compare the composition and age of thrombus collected at the site of coronary occlusion in patients with sudden death due to acute coronary artery occlusion and patients with an acute myocardial infarction without ventricular arrhythmia. The following hypothesis will be tested : fresh thrombus is more frequent in patients with sudden cardiac death versus patients with acute myocardial infarction without ventricular arrhythmia. Furthermore, coronary artery and systemic blood samples will be drawn in both groups and before coronary angioplasty procedures in patients with stable angina pectoris to determine the role of local and systemic inflammation and endothelial cell apoptosis in these settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sudden cardiac death without coronary artery occlusion
* Patients with acute myocardial infarction due to coronary artery occlusion
* Patients with stable angina treated with coronary angioplasty
* Written informed consent
* Social security

Exclusion Criteria:

* Pregnancy
* Small arteries that preclude the use of aspiration devices
* Sudden death without coronary lesions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2008-08; Primary Completion 2012-04 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Age of thrombus collected at the site of acute coronary occlusion. | one day

SECONDARY OUTCOMES:
Local and systemic inflammation and endothelial cell apoptosis in patients with sudden death due to acute coronary occlusion, acute myocardial infarction and stable angina treated with coronary angioplasty. | one day

CONTACTS AND LOCATIONS:
Overall Officials: Xavier JOUVEN, MD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Hopital Cochin, Paris, France